CLINICAL TRIAL: NCT03240250
Title: Randomized Study on Effects of Uniportal VATS Versus Triportal VATS for the Treatment of Stage I-II NSCLC
Brief Title: Randomized Study on Effects of Uniportal VATS Versus Triportal VATS
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 3564
Record Dates: First submitted 2017-07-13; First posted 2017-08-07 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2017-08

CONDITIONS: Lung Cancer
Keywords: VATS; Pulmonary lobectomy; Uniportal; Postoperative pain; Thoracic surgery
MeSH Terms: conditions — Lung Neoplasms; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uni-portal VATS: VATS uni-portal lobectomy and lymphoadenectomy
  Interventions: Procedure: VATS uni-portal lobectomy and lymphoadenectomy
- Three-portal VATS: VATS three-portal lobectomy and lymphoadenectomy
  Interventions: Procedure: VATS three-portal lobectomy and lymphoadenectomy

INTERVENTIONS:
Procedure: VATS uni-portal lobectomy and lymphoadenectomy — VATS uni-portal lobectomy and lymphoadenectomy
  Groups: Uni-portal VATS
Procedure: VATS three-portal lobectomy and lymphoadenectomy — VATS three-portal lobectomy and lymphoadenectomy, Copenhagen approach
  Groups: Three-portal VATS

SUMMARY:
For the treatment of stage I-II NSCLC, two mini-invasive techniques are mostly utilized: uni-portal and three-portal VATS. In the uniportal approach, the injury on a single intercostal space could determine a lower level of pain than the three-portal approach, allowing a better postoperative course. Few studies in Literature compare these techniques, and most of them are retrospective.

The main purpose of this randomized study is to compare uni-portal VATS with three-portal VATS, in terms of postoperative pain.

Secondary objectives of the study are valutations of:

* respiratory and functional capacity between the two groups
* operative time
* number of resected lymphnodes
* intra and postoperative complications, such as conversions to open surgery, amount of bleeding, prolonged air leaks, surgical site infections, pulmonary complications.

DETAILED DESCRIPTION:
Randomized cohort clinical trial, prospectic, monocentric. Procedure of randomization: the day before the operation, with the "Random Allocation Rule" technique

Arm 1: pulmonary lobectomy and lymphoadenectomy with uni-portal VATS approach

Arm 2: pulmonary lobectomy and lymphoadenectomy with three-portal VATS approach

Misurations Total analgesic consumption, normalized to morphine milligrams, recorded in the 7 days following the operation.

The choice of cumulative analgesic consumption as parameter of primary outcome is because pain valuation with VAS is significantly affected by individual variability.

Secondary outcomes: measure of postoperative pain with NRS at 2,6,12,24 hours and at 2,3,4,5,30 days from sugery. A pain score will be assigned to each patient after the total amount of NRS.

Respiratory function will be valuated with spirometry after 7 and 30 days from surgery, and compared with pre-operative tests.

All intraoperative parameters will be compared between the two groups: operative time (skin to skin), proportion of conversions to open surgery, number of resected lymphnodes, amount of bleeding.

Postoperative complications will be analyzed: rate of prolonged air leaks, surgical site infections, cardiac rythhm disfunctions, pulmonary complications, post-thoracotomy syndrome, as well as lenght of stay at the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cT1-2N0-1M0 NSCLC, maximum diameter 5cm
* ASA (American Society of Anestesiology) score 1-2-3

Exclusion Criteria:

* N2-N3 disease
* Induction chemotherapy
* Thoracic wall infiltration
* Previous thoracic surgery
* Important pleural adhesions
* Severe COPD, asthma, interstitial lung disease - Liver, kidney or cardiac failure
* Clotting disorders
* Analgesic allergy
* Sublobar resection, sleeve lobectomy, pneumonectomy
* Chronic analgesic, oppioids or cortisonic use
* Absence of informed consent

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical diagnosis of NSCLC, stage I-II, age 30-75, who undergo pulmonary lobectomy and limphadenectomy with radical intent
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-03-12 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Measurement of postoperative pain after uni-portal and three-portal VATS | 7 days
  Total analgesic consumption, normalized to morphine milligrams, recorded in the 7 days following the operation.

SECONDARY OUTCOMES:
Measure of postoperative pain with NRS at 2,6,12,24 hours and at 2,3,4,5,30 days from sugery. | 30 days
  A pain score will be assigned to each patient after the total amount of NRS
Valuation of respiratory function | 30 days
  Spirometry after 7 and 30 days from surgery, compared with pre-operative tests
Intraoperative parameters | 1 day
  Operative time (skin to skin, minutes)
Intraoperative bleeding | 1 day
  Amount of bleeding
Postoperative air leakage | 15 days
  Rate of prolonged air leaks
Postoperative complications | 1 month
  Cardiac rythhm disfunctions

CONTACTS AND LOCATIONS:
Overall Officials: Davide Tosi, Principal Investigator — Fondazione Ca' Granda IRCCS Policlinico Milan
Locations (1):
- Thoracic Surgery Unit - Fondazione IRCCS Ca' Granda Policlinico, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mendogni P, Mazzucco A, Palleschi A, Rosso L, Righi I, Carrinola R, Damarco F, Privitera E, Fumagalli J, Bonitta G, Nosotti M, Tosi D. Uniportal and three-portal video-assisted thoracic surgery pulmonary lobectomy for early-stage lung cancer (UNIT trial): study protocol of a single-center randomized trial. Trials. 2021 Feb 25;22(1):163. doi: 10.1186/s13063-021-05115-w. PMID 33632284